CLINICAL TRIAL: NCT05397717
Title: Prospective Study on Clinical Outcomes of Spontaneous Pneumothorax
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Doctor, Chinese University of Hong Kong
Other Study IDs: PTX_outcomes_prospective
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pneumothorax, Spontaneous
Keywords: Spontaneous pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spontaneous pneumothorax: A. Inclusion criteria i. All patients with a confirmed diagnosis of spontaneous pneumothorax on admission or during the hospital stay ii. Age greater than 18 years old iii. Chinese ethnicity iv. Able to sign written informed consent to participate in the study B. Exclusion criteria i. Pneumothorax was not found by thoracic imaging ii. Traumatic pneumothorax (including iatrogenic pneumothorax) iii. Pneumothorax with recent (within one month) lung resection surgery, that may be due to staple line issues iv. Trapped lung or non-expandable lungs, without evidence of air leakage v. Patients with psychiatric disease or cognitive impairment that may limit their ability of understanding or giving consent to the study
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — Observational, without interfering the patient care of treating doctors

SUMMARY:
Pneumothorax can be fatal if treatment is delayed or the pneumothorax is refractory. However, the mortality rates and their risk factors were mainly reported from retrospective studies, and local data regarding the mortality of spontaneous pneumothorax is scarce. This study aims at evaluating the in-hospital mortality and relevant clinical outcomes of spontaneous pneumothorax and identifying their predictive factors. The data collected from this study will also guide the planning of subsequent research to overcome the knowledge and service gap in managing spontaneous pneumothorax.

DETAILED DESCRIPTION:
Pneumothorax is a common respiratory disease and potentially recurrent, especially among patients with pre-existing lung diseases. It frequently requires in-patient care due to the need for invasive therapeutic procedures.

Pneumothorax can be fatal if treatment is delayed or the pneumothorax is refractory. The in-hospital mortality rate of spontaneous pneumothorax ranges between 0.7% and 15%, which is dependent on age, mode of admission and presence of co-existing lung diseases. However, the mortality rates and their risk factors were mainly reported from retrospective studies, and local data regarding the mortality of spontaneous pneumothorax is scarce. A multicentre retrospective study in Hong Kong evaluating patients admitted for pneumothorax in the year 2004 reported a mortality rate of 0.6% in those who had failed drainage with intercostal tube drainage. However, this study was not powered to investigate the overall mortality rate of pneumothorax and its predictive factor.

The majority of patients with pneumothorax can be discharged after the resolution of pneumothorax. However, a significant proportion of them may experience prolonged stay in the hospital due to various complications secondary to pneumothorax, including subcutaneous emphysema, persistent air leakage, and hospital-acquired pneumonia. All these conditions may cast negative impact on the overall prognosis, burden of pleural intervention and length of stay. Again, the incidence rate and determining factors of these conditions are seldomly reported.

This study aims at evaluating the in-hospital mortality and relevant clinical outcomes of spontaneous pneumothorax and identifying their predictive factors. The data collected from this study will also guide the planning of subsequent research to overcome the knowledge and service gap in managing spontaneous pneumothorax.

ELIGIBILITY:
Inclusion criteria

* All patients with a confirmed diagnosis of spontaneous pneumothorax on admission or during the hospital stay
* Age greater than 18 years old
* Chinese ethnicity
* Able to sign written informed consent to participate in the study

Exclusion criteria

* Pneumothorax was not found by thoracic imaging
* Traumatic pneumothorax (including iatrogenic pneumothorax)
* Pneumothorax with recent (within one month) lung resection surgery, that may be due to staple line issues
* Trapped lung or non-expandable lungs, without evidence of air leakage
* Patients with psychiatric disease or cognitive impairment that may limit their ability of understanding or giving consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spontaneous, both primary and secondary, pneumothorax, excluding traumatic causes
Sampling Method: Non-Probability Sample
Enrollment: 349 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the in-hospital mortality of spontaneous pneumothorax who admitted to the hospital | 36 months
  To evaluate the in-hospital mortality of spontaneous pneumothorax who admitted to the hospital

SECONDARY OUTCOMES:
To evaluate clinical characteristics and causes of pneumothorax | 36 months
  which include symptomatology, radiographical changes and presence of underlying chronic lung disease (that help ot classify the type of pneumothorax)
To evaluate the risk factors and causes for in-hospital mortality of spontaneous pneumothorax | 36 months
  which include age, body weight, extent of pneumothorax, number of pleural intervention and occurrence of complications
To evaluate other short and long-term outcomes due to pneumothorax | 36 months
  which include Occurrence of respiratory and non-respiratory complications secondary to pneumothorax, 30-day and 90-day mortality rates, length of hospital stay, readmission and recurrence rates

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No